CLINICAL TRIAL: NCT00379808
Title: Role of the Arachidonate 5-Lipoxygenase Pathway in Coronary Heart Disease
Brief Title: Study of the Arachidonate 5-Lipoxygenase Enzyme in Affecting the Risk for Coronary Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 06011312; AHA0615253B (Other Grant/Funding Number: American Heart Associatino)
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Results first posted 2012-07-23 (Estimated); Last update posted 2012-07-23 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Heart Disease
Keywords: coronary heart disease; montelukast; inflammation
MeSH Terms: conditions — Coronary Disease; Inflammation | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 1 lactose-containing capsule daily for 1 month
  Interventions: Drug: Placebo
- Montelukast 10 mg (Active Comparator): 1 montelukast 10 mg tablet (masked by capsule) daily for 1 month
  Interventions: Drug: montelukast

INTERVENTIONS:
Drug: montelukast — 10 mg tablet (masked by capsule) daily for 1 month
  Other Names: Singulair
  Arms: Montelukast 10 mg
Drug: Placebo — 1 lactose-containing capsule daily for 1 month
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a particular substance involved in inflammation, called leukotrienes, is involved in causing heart disease to occur or to progress.

DETAILED DESCRIPTION:
The focus of this study is to better understand why some adults develop heart disease and others do not. There are many known factors which play a role in causing heart disease, such as diet and lifestyle. Also, we know that inflammation, a process in the body which causes painful joints in arthritis or swelling at a site if injury, also contributes to heart disease. In particular, we will address whether leukotrienes, a component of inflammation, is involved in promoting heart disease. We will study this by giving subjects at high risk for heart disease a drug called montelukast which causes leukotrienes to have a reduced effect in the body. In addition for comparison, we will give other subjects a placebo for the same amount of time. These subjects will then be crossed-over and will receive either montelukast or placebo depending on which treatment they received first. We will compare these subjects using blood tests to see if subjects who take montelukast show signs of less inflammation caused by early heart disease as compared to subjects who do not.

ELIGIBILITY:
Inclusion Criteria:

-Current hypertension (blood pressure > 140/90 mmHg) or current use of anti-hypertensive medications AND

Exclusion Criteria:

* Current use of lipid-lowering medications
* Current use of montelukast
* Poorly controlled hypertension, where systolic blood pressure is greater than 160 or diastolic blood pressure is greater than 100
* Use of steroid drugs, non-steroidal anti-inflammatory drugs or other anti-inflammatory medications in the two weeks prior to enrollment. (low dose aspirin ( < 325 mg) is OK, but indication must be cardiovascular)
* Current recreational drug use
* Other cardiovascular disease or previous cardiovascular event. These include:
* history of angina pectoris
* history of heart failure
* presence of a cardiac pacemaker
* history of myocardial infarction
* previous revascularization procedure
* history cerebrovascular disease including stroke and transient ischemic attack
* Pregnancy or lactation
* Diabetes mellitus
* Lactose intolerance
* Contraindications to montelukast therapy
* Alcoholism
* Known hepatic disease
* Existing chronic obstructive pulmonary disease, asthma, allergic rhinitis
* Active chronic immune, infectious, neoplastic or inflammatory diseases requiring therapy (such as active Hepatitis B, Hepatitis C, human immunodeficiency virus (HIV))
* Immunosuppressant therapy or known immunosuppression due to disease high density lipoprotein (HDL) < 40 mg/dL (although this would be a risk factor for heart disease, because of preliminary data which indicates that montelukast may lower HDL levels, we will exclude patients with abnormally low HDL from study)
* Other criteria at investigator discretion that are deemed to make the subject a poor candidate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-07; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Johnson, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Family Practice Medical Group Clinic, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on flyers posted in public places, through recontact of patients in previous studies, and patients cared for in a family medicine clinic
Groups:
- Placebo Then Montelukast: Patients were randomized in a crossover design to placebo or montelukast. Patients int this randomization arm received 4 weeks of placebo then 4 weeks of montelukast. There was no washout between crossover
- Montelukast Then Placebo: Patients were randomized in a crossover design to placebo or montelukast. Patients in this arm got montelukast for 4 weeks and then placebo for 4 weeks. There was no washout period
Period: Intervention Period 1 (4 Weeks)
Arm/Group | Placebo Then Montelukast | Montelukast Then Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Intervention Period 2 (4 Weeks)
Arm/Group | Placebo Then Montelukast | Montelukast Then Placebo
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Patients were randomized in a crossover design, but baseline characteristics were presented for all participants. Likewise data are not separated by order of treatment because there were no order effects
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years]
  All study participants | 50.8 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: High-sensitivity C-reactive Protein
Description: measured in a CLIA clinical laboratory facility (Quest Diagnostics, Tampa, FL)
Time Frame: 1 month
Population: based on patients who completed the entire study
Measure: Median (Inter-Quartile Range); unit: mg/dl
Groups:
- Placebo: This is all participants who received placebo, whether in first or second intervention
- Montelukast: This is all patients who received montelukast, whether in the first or second intervention period
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
mg/dl | 1.0 [0.6 to 5.4] | 1.0 [0.5 to 8.3]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; Statistical power was calculated using G*Power (Dusseldorf, Germany). Based on previously observed effects of statin drugs on hsCRP levels, 22 subjects provided 80% power to detect a moderate effect on hsCRP levels; Test type: Superiority or Other; p = 0.22, Wilcoxon sign rank test; Median Difference (Net) = 0

2. Secondary Outcome: High Density Lipoprotein (HDL)-Cholesterol
Description: Lipid levels were determined at a clinical laboratory (Quest Diagnostics)
Time Frame: 1 month
Population: those completing entire study
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
mg/dl | 52 [46 to 68] | 50 [45 to 65]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; Null hypothesis is that montelukast does not affect HDL. Not powered for this endpoint; Test type: Superiority or Other; p = 0.57, Wilcoxon sign rank; percent difference = 3.8

3. Other Pre Specified Outcome: Triglycerides
Description: measured by a clinical laboratory; Quest Laboratories
Time Frame: 1 month
Population: those completing the entire study
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
mg/dl | 94 [75 to 129] | 104 [73 to 139]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; The null hypothesis is that montelukast does not affect triglycerides. The study was not powered to this outcome measure; Test type: Superiority or Other; p = 0.33, wilcoxon sign rank; percent difference = 7.4

4. Other Pre Specified Outcome: Monocyte Chemotactic Protein-1 (MCP-1)
Description: biomarker was measured by enzyme-linked immunosorbant assay (ELISA)
Time Frame: 1 month
Population: those who completed the entire study
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
pg/ml | 84 [72 to 105] | 94 [77 to 110]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; null hypothesis is that montelukast does not affect MCP-1. Study not powered to the biomarker; Test type: Superiority or Other; p = 0.12, Wilcoxon; percent difference = 11.9

5. Other Pre Specified Outcome: Interleukin 1 Receptor Antagonist (IL1ra)
Description: IL1ra was determined by enzyme-linked immunosorbant assay (ELISA)
Time Frame: 1 month
Population: all participants who completed the entire study
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
pg/ml | 518 [400 to 828] | 587 [429 to 1240]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; null hypothesis is that montelukast does not affect IL1ra; Test type: Superiority or Other; p = 0.03, wilcoxon sign rank test; percent difference = 13.3

6. Other Pre Specified Outcome: Epithelial Cell-derived Neutrophil-activating Peptide 78 (ENA-78)
Description: biomarker determined by enzyme-linked immunosorbant assay.
Time Frame: 1 month
Population: those completing the entire study
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Placebo | Montelukast
Number analyzed (Participants) | 21 | 21
pg/ml | 631 [441 to 1190] | 527 [175 to 1060]
Statistical Analysis 1: Comparison: Placebo vs Montelukast; null hypothesis is that montelukast does not affect ENA-78. The study is not powered to this biomarker; Test type: Superiority or Other; p = 0.09, wilcoxon sign rank; percent difference = 16.5

ADVERSE EVENTS:
Arm/Group | Placebo | Montelukast
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22

LIMITATIONS AND CAVEATS:
Because there were no order effects, the placebo groups were combined and the montelukast groups were combined. Therefore results from each of these are not reported by arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No